CLINICAL TRIAL: NCT01542047
Title: A Phase I Combination of Pazopanib and Carboplatin in Advanced Solid Malignancies
Brief Title: A Combination of Pazopanib and Carboplatin in Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low rate of accrual
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1015; PZP114405 (Other Grant/Funding Number: GlaxoSmithKline); NCI-2012-00915 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-02-06; First posted 2012-03-01 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Cancer, Metastatic
Keywords: Metastatic; Solid tumors; carboplatin; Paraplatin; Pazopanib; Votrient; Alkylating agent; Tyrosine kinase inhibitor; Metastatic disease
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Carboplatin; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin AUC5 + escalating pazopanib (Experimental): Carboplatin AUC5 IV Day 1 Pazopanib in escalating dosages, 200 mg to 800 mg starting on days 2 or 3 and ending on days 19 or 21
  Interventions: Drug: Carboplatin; Drug: Pazopanib

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be administered intravenously over approximately 30 minutes on day 1 of each cycle. The dosage used will be 5 AUC for the first 5 cycles, and will be increased to 6 AUC for the sixth cycle.
  Other Names: Paraplatin®; Paraplatin NovaPlus®
Drug: Pazopanib — Pazopanib will be administered orally at 200 to 800 mg/kg2. It will be given either on days 1 through 21 of each 3-week cycle, or if needed, it will be given on days 3 through 19.
  Other Names: Votrient

SUMMARY:
This study is designed to investigate the possibility that use of two similar but distinct drugs used together in treatment of advanced cancer might prove less toxic than either agent used alone, because dosages can be reduced for each agent. This is a phase I study that is designed to measure the frequency and levels of specific side effects when Carboplatin and Pazopanib are used in combination in advanced cancer patients. The possibility that anti-tumor activity will occur is also going to be investigated.

DETAILED DESCRIPTION:
Pazopanib has shown a promising anti-cancer activity as a single agent tyrosine kinase inhibitor. Activity against multiple tumors such as renal cell carcinoma (RCC) and neuroendocrine tumors have been documented, and it recently gained FDA approval for the treatment of metastatic kidney cancer. Also, an impressive activity as a single agent was recently reported in non-small cell lung cancer (NSCLC) in the neoadjuvant setting, where tumor shrinkage occurred in 86% of patients. Encouraging activity has also been seen in cervical cancer, ovarian cancer and soft tissue sarcomas. Multi-kinase targeting is an approach that may prove beneficial in a number of patient populations. In particular cancers such as breast, colon, pancreas etc., patients represent heterogeneous population of small groups based on genetic analyses. Some of these populations may benefit when multiple agents are given which have similar, but distinct targets of action. Dosages and therefore associated toxicities might be reduced by such an approach.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed advanced solid tumor type that is FDA approved for treatment with Carboplatin.
* Life expectancy at least 12 wks
* ECOG performance status of 0-2
* Provide written informed
* Adequate organ system function

FEMALES:

* Non-childbearing potential, who has had:
* A hysterectomy
* A bilateral oophorectomy (ovariectomy)
* A bilateral tubal ligation
* Is post-menopausal
* Complete abstinence from sexual intercourse 14 days before, during and at least 21 days after the last dose of investigational product
* Oral contraceptive
* Injectable progestogen
* Implants of levonorgestrel
* Estrogenic vaginal ring
* Percutaneous contraceptive patches
* Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
* Sole male partner sterilization prior to the female subject's entry - Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/ gel/ film/cream/suppository)
* If lactating: discontinue nursing prior to the first dose, during and for 14 days following the last dose of study drug

Exclusion Criteria:

* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug.
* Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:
* Active peptic ulcer disease
* Known intraluminal metastatic lesion/s with risk of bleeding
* Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or
* other gastrointestinal conditions with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:
* Malabsorption syndrome
* Major resection of the stomach or small bowel.
* Presence of uncontrolled infection
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula
* History of any one or more of the following cardiovascular conditions within the past 6 months:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Coronary artery bypass graft surgery
* Symptomatic peripheral vascular disease
* Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of greater than or equal to 140 mmHg or diastolic blood pressure (DBP) of greater than or equal to 90mmHg]

Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry.

* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major)
* Evidence of active bleeding or bleeding diathesis
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Hemoptysis within 8 weeks of first dose of study drug
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance with study procedures
* Treatment with any of the following anti-cancer therapies:
* Radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR
* Chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
* Any ongoing toxicity from prior anti-cancer therapy that is greater than Grade 1 and/or that is progressing in severity, except alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of Pazopanib when used in combination with Carboplatin | 3 months
  Patients will receive 200mg of Pazopanib, with later subjects receiving higher dosages up to 800mg of Pazopanib. If a given dose level is not well tolerated when given on all days (1-21) of each cycle, the study will no longer use that dosage. Later subjects may take Pazopanib from days 3-19 of the three week cycle to see if that dosing schedule is better tolerated.
  If patients experience side effects from Pazopanib or tests indicate some undesirable effects, then the dose level of Pazopanib that they are receiving may need to be adjusted, with increased monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Montasur Shaheen, MD, Principal Investigator — New Mexico Cancer Care Alliance/UNMCC
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: UNM Cancer Center — http://cancer.unm.edu/
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org